CLINICAL TRIAL: NCT05945953
Title: Comparison of Incentive Spirometer as a Visual Feedback Versus Deep Breathing Via Mirror Mediated Therapy on Pulmonary Function in Children With Spastic Cerebral Palsy
Brief Title: Incentive Spirometer as a Visual Feedback in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/01541 Ayesha Khalid
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy | interventions — Feedback, Sensory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentive spirometer as visual feedback (Experimental)
  Interventions: Other: Incentive spirometer as visual feedback
- Diaphragmatic breathing exercise (Mirror mediated therapy) (Active Comparator)
  Interventions: Other: Diaphragmatic breathing exercise (Mirror mediated therapy)

INTERVENTIONS:
Other: Incentive spirometer as visual feedback — Incentive spirometer as deep breathing then UE movement in sitting: Frequency: 2 sets of 10x Intensity: Up to tolerance (hold breath for 2-4 secs). Time: Twice a week Type: Deep breathing exercise UE movement: Gentle ROMs (5 reps)
  along with conventional Treatment; Passive stretching of spastic muscles, Strengthening of weak muscles using manual resistance, Diaphragmatic Breathing, Resisted Diaphragmatic Breathing (placing 5Ib sandbag on abdomen).
  Arms: Incentive spirometer as visual feedback
Other: Diaphragmatic breathing exercise (Mirror mediated therapy) — Diaphragmatic breathing exercise (Mirror mediated therapy): In front of mirror deep breathing with UE movement in sitting: Frequency: 1 cycle of 10x Intensity: Up to tolerance. Time: 3 times per week. Type: Deep breathing exercise. UE movement: Gentle ROMs (5 reps).
  along with conventional Treatment; Passive stretching of spastic muscles, Strengthening of weak muscles using manual resistance, Diaphragmatic Breathing, Resisted Diaphragmatic Breathing (placing 5Ib sandbag on abdomen).
  Arms: Diaphragmatic breathing exercise (Mirror mediated therapy)

SUMMARY:
Objective: To compare the effects of incentive spirometer as a visual feedback versus deep breathing via mirror mediated therapy on pulmonary function in children with spastic cerebral palsy. To determine the effects of incentive spirometer as a visual feedback versus deep breathing via mirror mediated therapy on sleep and quality of life in children with spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.
* Spastic diplegic, age above 5.
* According to modified Ashworth scale, moderate spasticity 1 to 3.
* Adequate cognition (will be assessed by using MMSE scale) in order to follow the instructions to use Incentive Spirometry and also able to comprehend single verbal command for breathing.
* Able to attend all sessions. (mentally and physically capable of attending session).
* Able to sit with support.

Exclusion Criteria:

* Participant falling in this category would be excluded of the study.
* Patients with any respiratory or cardiac disease that can affect their respiratory function.
* Patients with beta blockers or bronchodilators.
* Children with any cognitive impairment who are unable to follow instructions.
* Children with bone deformities, such as scoliosis or kyphosis.
* Children with any sort of auditory and visual defects.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 6 weeks
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 6 weeks
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters
Peak Expiratory Flow (PEF) | 6 weeks
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second

SECONDARY OUTCOMES:
Quality of life questionnaire for children (CPQOL-Child) | 6 weeks
  Changes from the baseline, This questionnaire has been specifically developed for children with cerebral palsy to measure the quality of life. Primary care giver questionnaire (4-12 years). These items can be recorded by the following formula: 1-2 (Very unhappy), 3-4(Unhappy), 5(neither happy nor unhappy), 6- 7(happy), 8-9 (very happy). If person scored 1, record to 0 If person scored 2, record to 12.5 If person scored 3, record to 25 If person scored 4, record to 37.5 If person scored 5, record to 50 If person scored 6, record to 62.5 If person scored 7, record to 75 If person scored 8, record to 87.5 If person scored 9, record to 100
Sleep (Sleep Disturbance Scale-SDSC) | 6 weeks
  This scale has been validated for children aged 6 to 15 years. The questionnaire is completed by caregiver or parents. It has internal consistency 0.71 to 0.79, test-retest reliability of 0.71 and diagnostic accuracy of 0.91. (32, 33) Scoring
  It is liker-type scale that indicates the following:
  1 means 'never' 5 means 'always' Total score (sum 6 factors' scores) Higher the score indicates more acute sleep disturbances. To obtain results, scores are tallied for each of six sleep disordere

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- NIRM (National Institute of Rehabilitation Medicine, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No